CLINICAL TRIAL: NCT02808091
Title: Phase II Trial of Bortezomib With Combination of Gemcitabine, Ifosfamide and Oxaliplatin (GIFOX-B)in Untreated NK/T Cell Lymphoma
Brief Title: Bortezomib With Combination of Gemcitabine, Ifosfamide and Oxaliplatin in Untreated NK/T Cell Lymphoma
Acronym: Gifox-B
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC1004
Record Dates: First submitted 2016-06-09; First posted 2016-06-21 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Extranodal NK-T-CELL LYMPHOMA
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early stage (IB or bulky disease - II) (Experimental): who will receive GIFOX-B chemotherapy followed by involved field radiotherapy.
  Interventions: Drug: GIFOX-Bortezomib; Radiation: IMRT
- Advanced stage (III - IV) (Experimental): will receive only chemotherapy alone
  Interventions: Drug: GIFOX-Bortezomib

INTERVENTIONS:
Drug: GIFOX-Bortezomib — GIFOX-Bortezomib will be given every 21 days for 4 cycles
  Arms: Early stage (IB or bulky disease - II)
Drug: GIFOX-Bortezomib — GIFOX-Bortezomib will be given every 21 days for a total of 6 cycles.
  Arms: Advanced stage (III - IV)
Radiation: IMRT — a minimum of 50 Gy of IMRT to tumor bed and neck (5 weeks)
  Other Names: Intensity-modulated radiation therapy
  Arms: Early stage (IB or bulky disease - II)

SUMMARY:
* Assess responses, progression free survival (PFS) and overall survival (OS) of the combination of GIFOX-B chemotherapy with intensity-modulated radiation therapy (IMRT) in Stage IB or bulky disease - II and without IMRT in Stage III - IV.
* Assess the toxicity and maximum tolerated dose of bortezomib administered in combination with GIFOX chemotherapy.

ELIGIBILITY:
Inclusion Criteria

1. Extranodal NK/T-cell lymphomas
2. Confirmed pathological diagnosis by the Department of Pathology SGH/NUH/TTSH.
3. Age more than or equals to 21 years.
4. Stages IB or bulky disease, II - IV
5. ECOG performance 0-2
6. Laboratory tests: ANC more than or equals to 1000/mm3, platelet more than or equals to 75,000/mm3. Creatinine less than or equals to 2x ULN or creatinine clearance more than or equals to 50 ml/min; AST and ALT less than or equals to 3x ULN. Total bilirubin < 1.5x ULN except < 3x ULN in patients with Gilbert's (as defined as > 80% unconjugated hyperbilirubinemia without other known cause); unless impairment is due to organ involvement by lymphoma.
7. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria

1. Had prior systemic chemotherapy. Patients may be entered if they have had prior limited-field radiotherapy or a short course of glucocorticoids or single agent chemotherapy for an urgent local problem at diagnosis (e.g. epidural cord compression, superior vena caval syndrome).
2. History of peripheral neuropathy
3. HIV positive
4. Presence of CNS disease
5. Hypersensitivity to bortezomib, boron, or mannitol
6. Contraindication to any cytotoxic drug contained in the chemotherapy regimen.
7. Female subject of child-bearing potential not willing to use an acceptable method of birth control (i.e. a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study and one year beyond treatment completion.
8. Female subject pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum β-human chorionic gonadotrophin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for women without child-bearing potential.
9. Invasive or active malignancy in past 2 years.
10. Serious concomitant medical illnesses that would jeopardize the patient's ability to receive the regimen with reasonable safety.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-03; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Response rates of bortezomib in combination with GIFOX (GIFOX-B) chemotherapy with or without intensity-modulated radiation therapy (IMRT) | 3 years
  Assess the response rates of bortezomib in combination with GIFOX (GIFOX-B) chemotherapy together with intensity-modulated radiation therapy (IMRT) in stage IB or bulky disease - II patients and chemotherapy alone in stage III - IV patients.

SECONDARY OUTCOMES:
Progression free survival (PFS) of the combination of GIFOX-B chemotherapy with IMRT in stage IB and III - IV patients | 3 years
Overall survival (OS) of the combination of GIFOX-B chemotherapy with IMRT in stage IB and III - IV patients | 5 years
Toxicity of bortezomib administered in combination with GIFOX chemotherapy | 3 years
  Access the toxicity of treatment according to CTC AE 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Soon Thye LIM, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre, Singapore, Singapore, Singapore